CLINICAL TRIAL: NCT03313635
Title: Prealbumin (Transthyretin) Levels in Men With Low-T
Brief Title: Evaluation of Prealbumin Levels in Men With Low-T
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AND-1-17
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Testosterone Deficiency
Keywords: Prealbumin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen serum samples are retained for this study and possible future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Men presenting with low-T: Men presenting with low-t will undergo a blood draw for evaluation of prealbumin levels.
  Interventions: Diagnostic Test: Men presenting with low-T

INTERVENTIONS:
Diagnostic Test: Men presenting with low-T — Evaluation of prealbumin levels.

SUMMARY:
This is a single-center study intended to evaluate prealbumin (transthyretin), a marker of anabolic metabolism, in men with androgen deficiency (Low-T). There is emerging evidence that prealbumin is an indicator of anabolic, versus catabolic, metabolism, and that lower levels may be associated with hypogonadism.

ELIGIBILITY:
Inclusion Criteria:

* Provide responses to standard questionnaires administered to subjects
* Written Informed Consent obtained
* Male sex at birth
* ≥ 40 and ≤ 75 years of age
* Presentation to the clinic with symptoms suggestive of low testosterone such as loss of libido, erectile dysfunction, cognitive or mood disturbances, etc.
* Able and willing to provide blood specimens and follow study schedule
* A final diagnosis can be established (androgen deficient versus not androgen deficient)

Exclusion Criteria:

* Previous exposure to exogenous T, DHEA, clomiphen citrate, or other Selective Estrogen Receptor Modulators, or OTC or herbals (Treatment Naïve)
* Use of opioid medication within 3 months prior to enrollment
* Serious psychiatric disease or uncontrolled medical illness, as suspected from medical history or clinical examination
* Use of any sex hormones or steroidal anabolic drug supplements (OTC or prescribed)(Treatment Naïve)
* Incapable of giving informed consent or complying with protocol or unwilling to comply with protocol requirements
* Diagnosis of prolactinoma

Ages: 40 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Male sex at birth
Study Population: Men between the ages of 40 and 75 presenting with signs/symptoms of low-T.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Prealbumin Levels | 1 day
  Evaluation of prealbumin levels in subjects presenting for evaluation of possible late onset adult hypogonadism diagnosed with and without Androgen Deficiency (AD)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Morgentaler, MD, Principal Investigator — Men's Health Boston
Locations (1):
- Men's Health Boston, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No